CLINICAL TRIAL: NCT06165133
Title: Task Shifting in InGuinal hErnia Repair Between Surgeons and Non-surgeon Physicians. A Multicentre Randomised Controlled Non-inferiority Trial.
Brief Title: Task Sharing in InGuinal hErnia Repair Between Surgeons and Non-surgeon Physicians
Acronym: TIGER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Ministry of Health, Ghana (Other Government); University of Abomey Calavi, Benin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RG_22-106
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Inguinal Hernia
Keywords: surgery; global surgery; inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: Multicentre, 2-arm, parallel group, assessor blinded, non-inferiority randomised controlled trial with an internal pilot.
Who Masked: Outcomes Assessor
Masking Description: The primary outcome assessment 90 days after surgery will be performed by a trained member of the research team who will not have access to the patient's hospital records or notes. If additional data needs to be retrospectively retrieved from hospital notes relating to a patient's secondary outcomes, then this may be accessed by any member of the research staff at that hospital (blinded or unblinded).
  The operating surgeon and patient are impossible to blind, as the patient will meet the surgeon on the day of surgery and introduce themselves. It is unethical and impractical not to tell a patient who is doing their surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Surgeon Physician (Experimental): The intervention arm is a mesh inguinal hernia repair performed by a non-surgeon physician (NSP). These are medical officers who have finished a 2-year mandatory house job. The medical officers will be trained to perform inguinal hernia repair by a certified surgical trainer in Ghana.
  Interventions: Other: Mesh inguinal hernia repair performed by Non-Surgeon Physicians (NSP)
- Control: Surgeon (Placebo Comparator): The control is a mesh inguinal hernia repair performed by a fully trained surgeon, defined as one who is accredited as fully trained with the Ghana College of Physicians and Surgeons, West African College of Surgeons, or equivalent. A trained surgeon will be assisted by an NSP who has completed the TIGER training programme. We anticipate that at least 5-10 fully trained surgeons will take part in the control arm.
  Interventions: Other: Mesh inguinal hernia repair performed by fully trained surgeons

INTERVENTIONS:
Other: Mesh inguinal hernia repair performed by Non-Surgeon Physicians (NSP) — Mesh inguinal hernia repair performed by Non-Surgeon Physicians (NSP) through an accredited training programme prior to commencing participation in the study
  Arms: Non-Surgeon Physician
Other: Mesh inguinal hernia repair performed by fully trained surgeons — Mesh inguinal hernia repair performed by fully trained surgeons, recognised by the Ghana College of Surgeons and Physicians and other recognised Surgical Colleges around the globe.
  Arms: Control: Surgeon

SUMMARY:
TIGER is a multicentre, 2-arm, parallel group, assessor blinded, non-inferiority randomised controlled trial with an internal pilot to assess if non-surgeon physicians (NSPs) can effectively perform mesh inguinal hernia repair compared to fully trained surgeons in adult patients with non-complicated inguinal hernia.

DETAILED DESCRIPTION:
Adult patients (18 years old to 60 years old, men and women) with non-complicated inguinal hernias suitable for elective repair will be recruited from at least 18 representative district hospitals in Low- and Middle-Income countries. Before and during a district hospital visit by a senior surgeon (at least once a year), a call will be made to the community, as is current practice (e.g., leaflet, radio, verbal at mosques, churches, market places, etc.).

Patients will attend the local district hospital on specific dates, which are contained within the announcement. A fully trained surgeon will examine the patient and identify patients according to the eligibility criteria, and if confirmed as eligible, they will be invited to enter the trial and consent obtained. If patients are not eligible for the trial, their care will follow the usual pathways.

After patient eligibility has been confirmed and informed consent has been obtained, patients will be randomised into the TIGER trial by a member of the TIGER research team at the site. Patients will be randomised to an operating list: NSP or surgeon list. The operating lists will be performed at the same hospital where the patient is randomised.

Patients are randomised to either of the following:

Intervention: Mesh inguinal hernia repair performed by Non-Surgeon Physicians (NSP) through an accredited training programme prior to commencing participation in the study.

Control: Mesh inguinal hernia repair performed by fully trained surgeons, recognised by the Ghana College of Surgeons and Physicians and other recognised Surgical Colleges around the globe.

A 'random element' will be included in the minimisation algorithm, so that each patient has a probability (unspecified here) of being randomised to a different intervention that they would have otherwise received.

Sample size: A sample size of 1782 patients (891 patients per arm) will be required to detect a non-inferiority margin of 2.5% in safe surgery, assuming a 90% baseline rate of safe surgery in the control arm (i.e., 10% of the patients are expected to have SSI or reoperation or recurrence in the control group). This allows for a 15% loss to follow-up, death before the primary outcome assessment, and misdiagnosis of inguinal hernia.

Inclusion Criteria

* Patients older than 18 years (male or female) and less or equal to 60 years (this criteria will be made country-specific. Each country will decide the lower and upper age limit for the trial),
* Primary inguinal hernia (unilateral) eligible for elective inguinal hernia repair
* Primary bilateral, but only one side being repaired
* Written informed consent of patient (signature or a fingerprint)

Exclusion Criteria

* Complex inguinal hernias: recurrent, obstructive, or femoral hernias
* Bilateral inguinal hernias undergoing simultaneous repair
* Inguinal hernias needing emergent surgical repair (e.g., incarcerated)
* Patient unable to complete post-operative follow-up

ELIGIBILITY:
Inclusion Criteria

* Patients older than <18 years> (male or female) and less or equal to 60 years
* Primary inguinal hernia (unilateral) eligible for elective inguinal hernia repair
* Primary bilateral, but only one side being repaired
* Written informed consent of patient (signature or a fingerprint)

Exclusion Criteria

* Complex inguinal hernias: recurrent, obstructive, or femoral hernias
* Bilateral inguinal hernias undergoing simultaneous repair
* Inguinal hernias needing emergent surgical repair (e.g., incarcerated)
* Patient unable to complete post-operative follow-up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1782 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety 90 days after surgery, defined by the absence of surgical site infection (SSI), reoperation or recurrence | 90 days post-op
  SSI will be defined as per CDC criteria within 90 days of inguinal hernia repair
  SSI after surgery will be defined according to CDC criteria. The following CDC definition will be used to identify deep incisional or superficial SSIs:
  Infection must occur within 30-days of the index operation AND Infection must involve the skin, subcutaneous, muscular or fascial layers of the incision AND
  Patient must have at least one of the following:
  Purulent drainage from the wound Organisms detected from a wound swab Wound opened spontaneously or by a clinician AND, at the surgical wound, the patient has at least one of: pain or tenderness; localised swelling; redness; heat; systemic fever (>38°C) Diagnosis of SSI by a clinician or radiological imaging Reoperation will be defined as any surgical complication requiring reoperation in theatre within 90 days of inguinal hernia repair.
  Recurrence will be defined as in the Reinforcement of Closure of Stoma Site (ROCSS) Trial.

SECONDARY OUTCOMES:
Surgical site infection | 30 and 90 days after surgery
  Surgical site infection at 30 days after surgery and 90 days after surgery (CDC criteria)
Reoperation | 30 and 90 days after surgery
  Reoperation at 30 days after surgery and 90 days after surgery (as described for the primary outcome)
Recurrence | 90 days and 1 year after surgery
  Inguinal hernia recurrence at 90 days after surgery and one year after surgery (as described for the primary outcome)
Quality of life (assessed using Abdominal Hernia-Q) | 1 year after surgery
  Quality of life at one year after surgery (using the Abdominal Hernia-Q questionnaire (AHQ)).
  (The AHQ is a validated patient reported outcome to assess hernia-specific quality of life in patients undergoing hernia operation. The pre-operative minimum score is 8 and post-operative is 16. The pre-operative maximum score is 32 and post-operative is 64; additional questions are asked after the operation relating to satisfaction around clinical care. Lower scores indicate a patient who is in greater pain/suffering greater disruption/dysphoria attributed to their hernia or dissatisfaction with their clinical care, high scores indicate the converse.
Chronic postoperative inguinal pain after surgery using the Faces Pain Scale - Revised (FPS-R) score | 90 days and 1 year after surgery
  Chronic postoperative inguinal pain 90 days and one year after surgery using FPS-R. This is from 0 - 10, with 0 indicating no pain, and 10 indicating extreme pain.
  A score of four or more (out of ten) will be used to define chronic pain in TIGER trial.
Postoperative inguinal pain after surgery using the Faces Pain Scale - Revised (FPS-R) score | 30 days after surgery
  Postoperative inguinal pain at 30 days after surgery (using the Faces Pain Scale - Revised (FPS-R) score). This is from 0 - 10, with 0 indicating no pain, and 10 indicating extreme pain.
  A higher score would signify a worse outcome for the patient.
Mortality | Within 30 days after surgery
  Mortality within 30 days of surgery
Duration of surgery | Measured intraoperatively
  Duration of surgery (in minutes)
Senior assistance during the surgical procedure. | Measured intraoperatively
  Senior assistance during the surgical procedure. For every patient operated on, it will be recorded if the professional performing the operation (surgeon or NSP) required assistance from a senior surgeon during the procedure. This is extremely relevant to measure as it will inform trial applicability in a real-world clinical scenario, particularly in the NSP arm but also in the surgeon arm.
Costs of all treatment | 30 days after surgery
  Cost-effectiveness 30 days after surgery. Resource use data will be collected as part of the economic evaluation of the two arms of the trial.
  The cost of mesh will be controlled across the trial. Intraoperative costs will be collected via a CRF for each operation. A hospital resource use CRF will be administered to patients at discharge to collect inpatient resource use. A resource use CRF administered to a patient at follow-up will be used to collect information on post-discharge costs. All resource use will be valued in monetary terms using unit costs/ prices where possible. Information on the costs of an inguinal hernia repair operation using a surgeon and NSP will be presented to decision makers to help set appropriate reimbursement levels for hospitals undertaking inguinal hernia repair.

CONTACTS AND LOCATIONS:
Overall Officials: Aneel Bhangu, Principal Investigator — University of Birmingham

IPD SHARING:
Plan to Share IPD: No
Hospital-level data will not be released or published. Country-level analyses will only be conducted with permission of lead investigators from each participating country. Local investigators may access their data across their country to perform country-level analyses (all participating hospitals should consent to their data being used in this way).